CLINICAL TRIAL: NCT06367751
Title: Implementation of Liquid Biopsies During Routine Clinical Care in Patients With Advanced Malignancies (LIQPLAT)
Acronym: LIQPLAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Research Center for Clinical Neuroimmunology and Neuroscience Basel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-00358; th23Kasenda
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor
Keywords: ctDNA

STUDY DESIGN:
Intervention Model Description: This is a trial using routinely collected health care data from an ongoing registry (AO_2023-00091) in cancer patients with advanced solid malignancies receiving first line systemic anti-cancer treatment for advanced disease. All patients will receive routine diagnostics, treatment and follow-up. All patients with a new cancer diagnosis will be assessed for eligibility based on the routinely collected information available in the registry. We will then randomly decide which eligible patients are invited to participate in the trial. If patients accept the invitation and intend to get a measurement of ctDNA, they have to provide written informed consent. The study comprises an external comparator arm with 75 (anticipated) cancer patients, and an active comparator arm with 150 (anticipated) cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Comparator (Experimental): Patients included in the ongoing registry AO_2023-00091.
  Patients will have ctDNA measurements being performed on blood samples collected as part of clinical routine.
  Interventions: Diagnostic Test: ctDNA measurement

INTERVENTIONS:
Diagnostic Test: ctDNA measurement — Blood samples are collected as part of standard of care and ctDNA measurements will be performed on these samples.

SUMMARY:
The goal of this study is to assess the implementation and feasibility of ctDNA measurements from blood samples obtained during routine clinical care of cancer patients in the University Hospital Basel.

Researchers will compare clinical and patient reported outcomes from the LIQPLAT study with patients who did not receive ctDNA measurements (external comparator from registry AO_2023-00091).

Blood samples will be drawn from the patients as part of routine care and ctDNA measurements will be performed on these samples.

DETAILED DESCRIPTION:
Liquid biopsies, in particular the analysis of circulating tumor DNA (ctDNA), have emerged as a promising tool for detecting and monitoring cancer. Measuring ctDNA in patients with solid malignancies may help to identify targetable alterations, measure disease burden, identify early mutations of resistance, tailor and deescalate cancer treatment, and predict patient prognosis. Although the adoption and application of ctDNA measurements for patients with solid tumors in routine clinical care is increasing, evidence supporting the integration of ctDNA into current practice is limited, especially for patients with advanced cancers.

This is a trial using routinely collected health care data from an ongoing registry (AO_2023-00091) in cancer patients with advanced solid malignancies receiving first line systemic anticancer treatment for advanced disease.

This trial will assess the feasibility and implementation of routine measurement of ctDNA and its association with clinical outcomes, including quality of life and survival. All patients will receive routine diagnostics, treatment and follow-up. All patients with a new cancer diagnosis will be assessed for eligibility based on the routinely collected information available in the registry. We will then randomly decide which eligible patients are invited to participate in the trial. If patients accept the invitation and intend to get a measurement of ctDNA, they have to provide written informed consent.

Results from ctDNA analyses will be discussed at the molecular tumor board, an established regular interdisciplinary meeting at the University Hospital Basel (part of routine care) to discuss patients with complex findings from tumor sequencing analyses. Treatment changes occurring during the trial duration will be at the discretion of treating physician and according to patient's preference as is routine standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a proven solid malignant disease, i.e. with solid malignant tumors where no primary surgical resection is planned OR solid malignant tumors that are locally advanced and inoperable OR solid tumors that are metastatic
* No prior treatment for advanced/metastatic disease
* Indication for medical anti-cancer treatment (including combined chemoradiotherapy) as judged by the treating physician
* Patient age 18 years and older
* General research consent of the University Hospital Basel

Exclusion Criteria:

● Patients with primary brain tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of patients in whom ctDNA was detectable before starting medical anticancer treatment | 1 time assessment at baseline
  Number and proportion of patients in whom ctDNA was detectable before starting medical anticancer treatment. Calculated as the number of patients with detectable ctDNA over the total number of patients included, expressed as a percentage.
Patients in whom actionable alterations were identified in ctDNA analysis | baseline, between month 2 and 3, between month 5 and 6, clinical event
  Patients in whom actionable alterations were identified in ctDNA analysis. Calculated as the number of patients with actionable alterations over the total number of patients included, expressed as a percentage.
  Clinical event is defined as suspicious or confirmed clinical or radiological disease progression or treatment discontinuation for any reason.
Turn-around time of ctDNA analysis | baseline, between month 2 and 3, between month 5 and 6, clinical event
  Time from ctDNA request until issuing the first report. Expressed as hours.
  Clinical event is defined as suspicious or confirmed clinical or radiological disease progression or treatment discontinuation for any reason.
ctDNA kinetics | up to 24 months
  Change in allelic frequency over time including relative changes from baseline.

SECONDARY OUTCOMES:
Number of ctDNA testing results that were successfully made available to the molecular tumor board | up to 24 months
  Number of ctDNA testing results that were successfully made available to the molecular tumor board.
Number of patients being positive for ctDNA and suspicious Clonal Hematopoiesis of Indeterminate Potential | up to 24 months
  Number of patients being positive for ctDNA and suspicious Clonal Hematopoiesis of Indeterminate Potential
Quality of life and physical function | month 3, month 6, month 12
  Global quality of life and physical function as measured by EORTC QLQ C30 and C15 (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire). Calculation of the scores follows the validated formulas as issued by the EORTC. Scores range from 0% to 100% for all domains with higher values representing better outcome.
Overall survival | up to 24 months
  Overall survival.
Survival rate 6 months | Month 6
  Survival rate 6 months.
Survival rate 12 months | Month 12
  Survival rate 12 months.
Time to next treatment line | up to 24 months
  Time to next treatment line, expressed in days.
Unplanned hospital admissions and emergency room visits | up to 24 months
  Number and proportion of unplanned hospital admissions and emergency room visits.
Progression free survival | up to 24 months
  Progression free survival as determined by routine imaging (e.g. CT scan, MRI), tumor marker (e.g. PSA). Defined as time from date of informed consent until disease progression or death, whatever occurs first.
Number of ctDNA analyses with a valid result | up to 24 months
  Number of ctDNA analyses with a valid result - that is all ctDNA analyses conducted without any observed technical errors.

OTHER OUTCOMES:
Patients being referred and recruited to a different interventional clinical trial | up to 24 months
  Number and proportion of patients being referred and recruited to a different interventional clinical trial.
Tissue biopsies per patient | up to 24 months
  Number of (solid) tissue biopsies per patient and proportion of patients receiving a biopsy.
Imaging per patient | up to 24 months
  Number of imaging per patient (CT, PET/CT or MRI).
Blood products per patient | up to 24 months
  Number of blood products per patient.
Cumulative doses of cancer drug treatments administered | up to 24 months
  Cumulative doses of cancer drug treatments administered.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kasenda, PD. Dr. med et Dr. phil., Principal Investigator — USB
Locations (1):
- Department of Medical Oncology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request following SPHN (https://sphn.ch/) guidelines for data sharing.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Schwenke JM, Schmitt AM, McLennan S, Janiaud P, Laubli H, Binder M, Alborelli I, Matter MS, Hinke J, Widmer CC, Hemkens LG, Kasenda B, Briel M. Mixed-methods process evaluation of ctDNA use to guide decision-making in patients with advanced solid cancers: study protocol for a substudy of the LIQPLAT trial. BMJ Open. 2025 Oct 28;15(10):e100537. doi: 10.1136/bmjopen-2025-100537. PMID 41151945